CLINICAL TRIAL: NCT02515292
Title: Multidimensional Modeling in Evaluation of Infants With Intrauterine Growth Restriction
Brief Title: Evaluation of Infants With Intrauterine Growth Restriction
Acronym: ModeInfIUGR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Hășmășanu Monica Gabriela, MD, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: 142 /181/ 20.05.2014
Record Dates: First submitted 2015-07-29; First posted 2015-08-04 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Intrauterine Growth Restriction
Keywords: IUGR (intrauterine growth restriction); IGF2 (insulin-like growth factor 2); morbidity
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- IUGR: newborn with intrauterine growth restriction: Inclusion criteria:
  * newborn infants with symmetrical (both weight and height lower than 10th percentile) or asymmetrical (birth weight is lower than 10th percentile but height and age-appropriated height) intrauterine growth restriction
  * agreement of the parents that their child to be included in the study
- control: newborn without intrauterine growth restriction: Inclusion criteria:
  - matches newborn without intrauterine growth restriction in terms of gender and gestational age as IUGR group

SUMMARY:
Purpose: Clinical assessment (anthropometric) and paraclinical (biochemical and immunological by dosing serum insuline growth factors IGF1 and IGF2 and their receptors) of neonates with intrauterine growth restriction (IUGR) and the integration in a multidimensional statistical model .

Objectives:

1. IGF1 and IGF2 evaluation of serum and IGF1 receptor, IGF2 receptor and IGF2 receptor gene expression in cord blood from newborns with intrauterine growth restriction (IUGR). (Prospective)
2. Evaluation and monitoring of anthropometric, clinical (non-cardiac morbidity) and paraclinical. (Retrospective & prospective)
3. Evaluation and monitoring of morphological and functional by echocardiography. (Prospective)
4. Integrating multidimensional clinical and paraclinical parameters in a statistical model for evaluating newborn with intrauterine growth restriction.

ELIGIBILITY:
Inclusion Criteria:

* newborns with intrauterine growth restriction (IUGR): weight below the 10th percentile for gestational age
* parental consent for enrollment

Exclusion Criteria:

* IUGR neonates in the context chromosomopathies: trisomy 21, trisomy 18.
* neonates with congenital heart disease
* twins
* refusal of parents for participation to the study

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Population with IUGR from a 3rd level maternity from Nord-West of Romania
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of serum IGF2 | baseline
  serum IGF2
Evaluation of IGF2 receptors | baseline
  serum IGF2 receptors

SECONDARY OUTCOMES:
Genetic evaluation | baseline
  Number of subjects homozygous (A or G) and heterozygous (A/G) using forward primer: 5'- CTTGGACTTTGAGTCAAATTGG-3' and reverse primer: 5'-GGTCGTGCCAATTACATTTCA-3' genetic expression of IGF2 receptors. The groups will be evaluated in regards of polymorphism and allele frequencies.
Clinical assessment | baseline
  Number of cases with respiratory distress, hyperbilirubinemia, early and late sepsis, hypoglicemia, necrozant enterocolitis or other co-morbidities.
Cardiac morphological and functional evaluation | baseline and follow-up (1 month and/or 6 months)
  Eco cardiac measurements will be performed to all participants and the morphological and functional data will be recorded baseline for all participant (IUGR and controls). As results number of subjects with cardiac morphological and functional evaluation will be according with subjects included in the study and those subjects with cardiac modification or those from case group will be evaluated dynamically.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Zaharie, PhD, MD, Study Chair — Iuliu Hațieganu Medicine and pharmacy University
Locations (1):
- Neonatal-Ward, 1st Gynecology Clinic, Cluj-Napoca, Cluj, Romania